CLINICAL TRIAL: NCT02786654
Title: β Blocker Use and Mortality in Hospital Survivors of Acute Myocardial Infarction Without Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Tatendashe Bernadette Dondo, Research assistant, University of Leeds
Other Study IDs: PG/13/81/30474BB
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; mortality; evidence-based care; Myocardial Ischaemia National Audit Project; β blockers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years

SUMMARY:
The aim of the study is to investigate the association between the use of β blockers and mortality among hospital survivors of acute myocardial infarction without heart failure.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction patients only
* aged 18 to 100 years

Exclusion Criteria:

* other final diagnosis besides acute myocardial infarction
* died in-hospital
* patients with missing mortality data
* aged > 100
* patients with previous acute myocardial infarction or angina
* patients who have received coronary interventions before
* patients with heart failure
* patients with β blocker prior use
* patients contraindicated for β blocker use
* patients with use of a loop diuretic

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised of 179,810 in hospital survivors of acute myocardial infarction without heart failure recorded in the Myocardial Ischaemia National Audit Project registry between 2007 and June 2013
Sampling Method: Non-Probability Sample
Enrollment: 179810 (Actual)
Dates: Start 2007-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1 year

SECONDARY OUTCOMES:
All cause mortality | 6 months
All cause mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris P Gale, FRCP, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dondo TB, Hall M, West RM, Jernberg T, Lindahl B, Bueno H, Danchin N, Deanfield JE, Hemingway H, Fox KAA, Timmis AD, Gale CP. beta-Blockers and Mortality After Acute Myocardial Infarction in Patients Without Heart Failure or Ventricular Dysfunction. J Am Coll Cardiol. 2017 Jun 6;69(22):2710-2720. doi: 10.1016/j.jacc.2017.03.578. PMID 28571635